CLINICAL TRIAL: NCT05987787
Title: Staple-line Suture Reinforcement: Could it Help Contain the Leak?
Brief Title: Suture Reinforcement to Reduce the Leak Rate After Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Giovanna Pavone, Medical doctor, University of Foggia
Other Study IDs: 8
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Leak, Anastomotic; Bleeding
MeSH Terms: conditions — Obesity, Morbid; Anastomotic Leak; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese patients underwent laparoscopic sleeve gastrectomy with suture reinforcement: Laparoscopic sleeve gastrectomy running seromuscular stitches at the proximal third of the stapled line using unidirectional 2/0 barbed sutures to invaginate the staple line completely.
  Interventions: Procedure: laparoscopic sleeve gastrectomy with suture reinforcement
- Obese patients underwent laparoscopic sleeve gastrectomy without suture reinforcement: Laparoscopic sleeve gastrectomy without staple line reinforcement.
  Interventions: Procedure: laparoscopic sleeve gastrectomy without suture reinforcement

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy without suture reinforcement — The procedure begins by dissecting the small branches of the gastroepiploic arch 6 cm from the pylorus. The dissection continues along the great curvature of the stomach, remaining very close to the gastric wall, up to the short gastric vessels which are also dissected. The stomach is then raised to expose its posterior wall and the adhesions are lysed. His angle is fully mobilized and the left diaphragmatic pillar exposed. The gastric tubule is created on the guide of a 40 F Bugie using mechanical suturing machines with charges of different thickness depending on the thickness of the gastric wall. At this point the bougie is removed and the resected stomach is extracted from the abdomen through the mesogastric access.
  Groups: Obese patients underwent laparoscopic sleeve gastrectomy without suture reinforcement
Procedure: laparoscopic sleeve gastrectomy with suture reinforcement — The procedure begins by dissecting the small branches of the gastroepiploic arch 6 cm from the pylorus. The dissection continues along the great curvature of the stomach, remaining very close to the gastric wall, up to the short gastric vessels which are also dissected. The stomach is then raised to expose its posterior wall and the adhesions are lysed. His angle is fully mobilized and the left diaphragmatic pillar exposed. The gastric tubule is created on the guide of a 40 F Bugie using mechanical suturing machines with charges of different thickness depending on the thickness of the gastric wall. At this point the bougie is removed and the resected stomach is extracted from the abdomen through the mesogastric access. At this point, it is applied running seromuscular stitches at the proximal third of the stapled line using unidirectional 2/0 barbed sutures to invaginate the staple line completely.
  Groups: Obese patients underwent laparoscopic sleeve gastrectomy with suture reinforcement

SUMMARY:
Staple line reinforcement (SLR) has been suggested as a mean of reducing the risk of sleeve leakage or bleeding. The aim of this study is to analyze if the suture reinforcement can be used to reduce the leakage rate after sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40 kg/m2
* BMI>35 kg/m2with at least one associated major comorbidity

Exclusion Criteria:

* secondary obesity due to endocrine and psychological disorders
* patients under antiaggregant and anticoagulant therapy
* re-do surgery.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Body mass index (BMI) ≥35-39 kg/m2 with one obesity- associated co-morbidity or BMI≥40kg/m2, age ≥ 18 years. Before surgery, patients underwent a standardized psychological and physical evaluation which includes blood chemistry tests, chest x-rays, electrocardiogram and cardiological examinations, nutritional evaluation, esophagogastroduodenoscopy, spirometry and psychiatric evaluation .
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
the importance of staple line reinforcement | 1 year
  reduction of the leak rate in the suture group
the importance of staple line reinforcement | During Surgery
  the differences of operative time between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT05987787/Prot_000.pdf